CLINICAL TRIAL: NCT00938639
Title: A Phase II, Single-centre, Randomised, Observer-blind Study to Evaluate the Immunogenicity, Safety and Tolerability of CSL's Monovalent H1N1 Influenza Virus Vaccine in Healthy Adults Aged 18 to < 65 Years.
Brief Title: A Clinical Trial of CSL's 2009 H1N1 Influenza Vaccine (CSL425) in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CSLCT-CAL-09-59
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Results first posted 2013-11-21 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-04

CONDITIONS: Influenza Caused by the Novel Influenza A (H1N1) Virus
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CSL425 (15 mcg) (Experimental): 15 mcg of haemagglutinin antigen per dose. 0.25 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21
  Interventions: Biological: CSL425
- CSL425 (30 mcg) (Experimental): 30 mcg of haemagglutinin antigen per dose. 0.5 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21
  Interventions: Biological: CSL425

INTERVENTIONS:
Biological: CSL425 — CSL's 2009 H1N1 Influenza Vaccine, thimerosal 0.01% (weight/volume)
  Arms: CSL425 (15 mcg)
Biological: CSL425 — CSL's 2009 H1N1 Influenza Vaccine, thimerosal 0.01% (weight/volume)
  Arms: CSL425 (30 mcg)

SUMMARY:
The purpose of the study is to determine whether CSL425 is a safe and effective vaccine for eliciting an immune response to H1N1 influenza in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged >= 18 to < 65 years at the time of providing informed consent.

Exclusion Criteria:

* Known hypersensitivity to a previous dose of influenza virus vaccine or allergy to eggs, chicken protein, thiomersal, neomycin, polymyxin, or any components of the Study Vaccine.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2009-07; Primary Completion 2009-09 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director, Vaccines Clinical Development, Study Director — Seqirus
Locations (1):
- Study Site, Adelaide, South Australia, Australia

REFERENCES:
- [Result] Greenberg ME, Lai MH, Hartel GF, Wichems CH, Gittleson C, Bennet J, Dawson G, Hu W, Leggio C, Washington D, Basser RL. Response to a monovalent 2009 influenza A (H1N1) vaccine. N Engl J Med. 2009 Dec 17;361(25):2405-13. doi: 10.1056/NEJMoa0907413. Epub 2009 Sep 10. PMID 19745216

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Started | 120 | 120
Completed | 117 | 116
Not Completed | 3 | 4
Not completed — Moved away from study area | 0 | 1
Not completed — Lost to Follow-up | 1 | 2
Not completed — Family issues | 1 | 1
Not completed — Participant noncompliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg) | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (15.12) | 42.9 (15.39) | 43.7 (15.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 67 | 134
  Male | 53 | 53 | 106

OUTCOME MEASURES:

1. Primary Outcome: Haemagglutination Inhibition (HI) and Microneutralisation (MN) Antibody Titre Seroconversion Rate After the First Vaccination
Description: Antibody titre seroconversion was defined as participants with a pre-vaccination titre of less than 1:10 achieving a post-vaccination antibody titre of 1:40 or more; or participants with a pre-vaccination titre of 1:10 or more achieving a four-fold or greater increase in post-vaccination HI titre.
Time Frame: Before and 21 days after the first vaccination
Population: The Evaluable Population (for the first vaccination) comprised all randomised participants who received the first study vaccination; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 119
percentage of participants
  Seroconversion rate - HI | 74.2 [65.4 to 81.7] | 81.5 [73.4 to 88.0]
  Seroconversion rate - MN | 77.5 [69.0 to 84.6] | 75.6 [66.9 to 83.0]

2. Primary Outcome: HI and MN Antibody Titre Seroconversion Rate After the Second Vaccination
Description: as for outcome 1
Time Frame: Before and 21 days after the second vaccination
Population: The Evaluable Population (for the second vaccination) comprised all randomised participants who received the second study vaccination; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 117 | 115
percentage of participants
  Seroconversion rate - HI | 82.1 [73.9 to 88.5] | 89.6 [82.5 to 94.5]
  Seroconversion rate - MN | 87.2 [79.7 to 92.6] | 83.5 [75.4 to 89.7]

3. Primary Outcome: Geometric Mean Fold Increase (GMFI) in the HI and MN Antibody Titre After the First Vaccination
Description: GMFI in antibody titre was defined as the geometric mean of the fold increase in the post-vaccination antibody titre over the pre-vaccination antibody titre.
Time Frame: Before and 21 days after the first vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold increase
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 119
geometric mean fold increase
  GMFI - HI | 11.83 [8.91 to 15.70] | 19.54 [14.58 to 26.20]
  GMFI - MN | 24.83 [17.56 to 35.11] | 39.70 [26.68 to 59.06]

4. Primary Outcome: GMFI in the HI and MN Antibody Titer After the Second Vaccination
Description: as for outcome 3
Time Frame: Before and 21 days after the second vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold increase
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 117 | 115
geometric mean fold increase
  GMFI - HI | 16.00 [12.36 to 20.71] | 23.30 [17.92 to 30.29]
  GMFI - MN | 32.30 [23.96 to 43.54] | 46.50 [32.83 to 65.87]

5. Primary Outcome: Percentage of Participants Achieving a HI or MN Antibody Titre of 1:40 or More After the First Vaccination
Time Frame: 21 days after the first vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 119
percentage of participants
  Participants with HI titer ≥ 1:40 | 95.0 [89.4 to 98.1] | 89.1 [82.0 to 94.1]
  Participants with MN titer ≥ 1:40 | 88.3 [81.2 to 93.5] | 83.2 [75.2 to 89.4]

6. Primary Outcome: Percentage of Participants Achieving a HI or MN Antibody Titre of 1:40 or More After the Second Vaccination
Time Frame: 21 days after the second vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 117 | 115
percentage of participants
  Participants with HI titer ≥ 1:40 | 98.3 [94.0 to 99.8] | 96.5 [91.3 to 99.0]
  Participants with MN titer ≥ 1:40 | 95.7 [90.3 to 98.6] | 92.2 [85.7 to 96.4]

7. Secondary Outcome: HI and MN Antibody Titre Seroconversion Rate After the First Vaccination by Age Group
Description: Antibody titre seroconversion was defined as participants with a pre-vaccination titre of less than 1:10 achieving a post-vaccination antibody titre of 1:40 or more; or participants with a pre-vaccination titre of 1:10 or more achieving a four-fold or greater increase in post-vaccination HI titre.
  Adults were aged from 18 to 49 years; Older adults were aged from 50 to 64 years.
Time Frame: Before and 21 days after the first vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- CSL425 (15 mcg), Adult; CSL425 (15 mcg), Older Adult: 15 mcg of haemagglutinin antigen per dose. 0.25 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21
- CSL425 (30 mcg), Adult; CSL425 (30 mcg), Older Adult: 30 mcg of haemagglutinin antigen per dose. 0.5 mL intramuscular injection into the deltoid region of the arm on Day 0 and Day 21
Arm/Group | CSL425 (15 mcg), Adult | CSL425 (15 mcg), Older Adult | CSL425 (30 mcg), Adult | CSL425 (30 mcg), Older Adult
Number analyzed (Participants) | 58 | 62 | 61 | 58
percentage of participants
  Seroconversion rate - HI | 77.6 [64.7 to 87.5] | 71.0 [58.1 to 81.8] | 85.2 [73.8 to 93.0] | 77.6 [64.7 to 87.5]
  Seroconversion rate - MN | 82.8 [70.6 to 91.4] | 72.6 [59.8 to 83.1] | 83.6 [71.9 to 91.8] | 67.2 [53.7 to 79.0]

8. Secondary Outcome: HI and MN Antibody Titre Seroconversion Rate After the Second Vaccination by Age Group
Description: as for outcome 7
Time Frame: Before and 21 days after the second vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg), Adult | CSL425 (15 mcg), Older Adult | CSL425 (30 mcg), Adult | CSL425 (30 mcg), Older Adult
Number analyzed (Participants) | 55 | 62 | 58 | 57
percentage of participants
  Seroconversion rate - HI | 83.6 [71.2 to 92.2] | 80.6 [68.6 to 89.6] | 87.9 [76.7 to 95.0] | 91.2 [80.7 to 97.1]
  Seroconversion rate - MN | 89.1 [77.8 to 95.9] | 85.5 [74.2 to 93.1] | 86.2 [74.6 to 93.9] | 80.7 [68.1 to 90.0]

9. Secondary Outcome: GMFI in the HI and MN Antibody Titre After the First Vaccination by Age Group
Description: GMFI in antibody titre was defined as the geometric mean of the fold increase in the post-vaccination antibody titre over the pre-vaccination antibody titre.
  Adults were aged from 18 to 49 years; Older adults were aged from 50 to 64 years.
Time Frame: Before and 21 days after the first vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold increase
Arm/Group | CSL425 (15 mcg), Adult | CSL425 (15 mcg), Older Adult | CSL425 (30 mcg), Adult | CSL425 (30 mcg), Older Adult
Number analyzed (Participants) | 58 | 62 | 61 | 58
geometric mean fold increase
  GMFI - HI | 15.13 [9.97 to 22.96] | 9.39 [6.37 to 13.84] | 25.79 [17.00 to 39.11] | 14.60 [9.68 to 22.02]
  GMFI - MN | 36.73 [22.23 to 60.68] | 17.21 [10.72 to 27.64] | 54.91 [31.75 to 94.96] | 28.22 [15.80 to 50.41]

10. Secondary Outcome: GMFI in the HI and MN Antibody Titre After the Second Vaccination by Age Group
Description: as for outcome 9
Time Frame: Before and 21 days after the second vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold increase
Arm/Group | CSL425 (15 mcg), Adult | CSL425 (15 mcg), Older Adult | CSL425 (30 mcg), Adult | CSL425 (30 mcg), Older Adult
Number analyzed (Participants) | 55 | 62 | 58 | 57
geometric mean fold increase
  GMFI - HI | 18.00 [12.17 to 26.62] | 14.41 [10.16 to 20.45] | 26.01 [17.69 to 38.25] | 20.82 [14.44 to 30.02]
  GMFI - MN | 37.95 [23.39 to 61.58] | 28.00 [19.26 to 40.70] | 55.79 [33.51 to 92.90] | 38.63 [23.79 to 62.73]

11. Secondary Outcome: Percentage of Participants Achieving a HI or MN Antibody Titre of 1:40 or More After the First Vaccination by Age Group
Description: Adults were aged from 18 to 49 years; Older adults were aged from 50 to 64 years.
Time Frame: 21 days after the first vaccination
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg), Adult | CSL425 (15 mcg), Older Adult | CSL425 (30 mcg), Adult | CSL425 (30 mcg), Older Adult
Number analyzed (Participants) | 58 | 62 | 61 | 58
percentage of participants
  Participants with HI titer ≥ 1:40 | 96.6 [88.1 to 99.6] | 93.5 [84.3 to 98.2] | 98.4 [91.2 to 100.0] | 79.3 [66.6 to 88.8]
  Participants with MN titer ≥ 1:40 | 94.8 [85.6 to 98.9] | 82.3 [70.5 to 90.8] | 95.1 [86.3 to 99.0] | 70.7 [57.3 to 81.9]

12. Secondary Outcome: Percentage of Participants Achieving a HI or MN Antibody Titre of 1:40 or More After the Second Vaccination by Age Group
Description: Adults were aged from 18 to 49 years; Older adults were aged from 50 to 64 years.
Time Frame: 21 days after the second vaccination
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg), Adult | CSL425 (15 mcg), Older Adult | CSL425 (30 mcg), Adult | CSL425 (30 mcg), Older Adult
Number analyzed (Participants) | 55 | 62 | 58 | 57
percentage of participants
  Participants with HI titer ≥ 1:40 | 98.2 [90.3 to 100.0] | 98.4 [91.3 to 100.0] | 100.0 [93.8 to 100.0] | 93.0 [83.0 to 98.1]
  Participants with MN titer ≥ 1:40 | 100.0 [93.5 to 100.0] | 91.9 [82.2 to 97.3] | 100.0 [93.8 to 100.0] | 84.2 [72.1 to 92.5]

13. Secondary Outcome: Percentage of Participants With a Baseline Titre Less Than 1:10 Achieving Seroconversion After Vaccination
Description: The number of participants with a baseline titre less than 1:10 differed according to antibody assay (HI or MN) and is shown in the category titles accordingly. The total number of participants analysed includes all evaluable participants; however, the analysis is stratified by baseline titre and those participants with a baseline titre less than 1:10 are presented in this outcome measure while those with a baseline titre of 1:10 or more are presented in a separate outcome measure.
  Antibody titre seroconversion was defined as participants with a pre-vaccination titre of less than 1:10 achieving a post-vaccination titre of 1:40 or more; or participants with a pre-vaccination titre of 1:10 or more achieving a four-fold or greater increase in post-vaccination HI titre.
Time Frame: Before and 21 days after each vaccination
Population: The Evaluable Population comprised all randomised participants who received the first (or second, as appropriate) study vaccination; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 119
percentage of participants
  After the first vaccination - HI (N = 42, 49) | 92.9 [80.5 to 98.5] | 83.7 [70.3 to 92.7]
  After the second vaccination - HI (N = 42, 47) | 95.2 [83.8 to 99.4] | 93.6 [82.5 to 98.7]
  After the first vaccination - MN (N = 62, 73) | 77.4 [65.0 to 87.1] | 74.0 [62.4 to 83.5]
  After the second vaccination - MN (N = 60, 71) | 91.7 [81.6 to 97.2] | 87.3 [77.3 to 94.0]

14. Secondary Outcome: Percentage of Participants With a Baseline Titre Greater Than or Equal to 1:10 Achieving Seroconversion After Vaccination
Description: The number of participants with a baseline titre greater than or equal to 1:10 differed according to antibody assay (HI or MN) and is shown in the category titles accordingly. The total number of participants analysed includes all evaluable participants; however, the analysis is stratified by baseline titre and those participants with a baseline titre of 1:10 or more are presented in this outcome measure while those with a baseline titre less than 1:10 are presented in a separate outcome measure.
  Antibody titre seroconversion was defined as participants with a pre-vaccination titre of less than 1:10 achieving a post-vaccination titre of 1:40 or more; or participants with a pre-vaccination titre of 1:10 or more achieving a four-fold or greater increase in post-vaccination HI titre (ie, a significant increase in antibody titre after vaccination).
Time Frame: Before and 21 days after each vaccination
Population: The Evaluable Population comprised all randomised participants who received the study vaccination; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 119
percentage of participants
  After the first vaccination - HI (N = 78, 70) | 64.1 [52.4 to 74.7] | 80.0 [68.7 to 88.6]
  After the second vaccination - HI (N = 75, 68) | 74.7 [63.3 to 84.0] | 86.8 [76.4 to 93.8]
  After the first vaccination - MN (N = 58, 46) | 77.6 [64.7 to 87.5] | 78.3 [63.6 to 89.1]
  After the second vaccination - MN (N = 57, 44) | 82.5 [70.1 to 91.3] | 77.3 [62.2 to 88.5]

15. Secondary Outcome: GMFI in the HI Antibody Titre 180 Days After the Second Vaccination
Description: The GMFI in antibody titre was calculated by taking the anti-logs of the means of the log transformed fold-increases in the antibody titre 180 days after the second vaccination over the antibody titre 21 days after the second vaccination.
Time Frame: 21 days and 180 days after the second vaccination
Population: The Evaluable Population comprised all randomised participants who received the second study vaccination; provided both pre- and post-vaccination blood samples; were not excluded from analyses (eg, for the use of a prohibited medication or a laboratory-confirmed 2009 H1N1 infection between Visit 1 and Visit 3).
Measure: Geometric Mean (95% Confidence Interval); unit: geometric mean fold increase
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 115 | 111
geometric mean fold increase | 0.49 [0.44 to 0.55] | 0.42 [0.38 to 0.47]

16. Secondary Outcome: Percentage of Participants Achieving a HI Antibody Titre of 1:40 or More 180 Days After the Second Vaccination
Time Frame: 180 days after the second vaccination
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 115 | 111
percentage of participants | 95.7 [90.1 to 98.6] | 91.9 [85.2 to 96.2]

17. Secondary Outcome: Frequency and Intensity of Solicited Local Adverse Events (AEs) After the First Vaccination
Description: Solicited AEs included AEs that were specifically sought for. Grade 3 solicited AE definitions: Prevented normal daily activities; Size > 100 mm for injection site redness, induration/swelling, and bruising.
Time Frame: From Day 0 to Day 6 after the first vaccination
Population: The Safety Population comprised all participants who received at least one dose of the vaccine and provided follow-up safety data.
Measure: Number; unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 120
percentage of participants
  Any local solicited AE | 40.0 | 49.2
  Any pain at injection site | 20.8 | 22.5
  Grade 3 pain at injection site | 0 | 0
  Any redness at injection site | 0.8 | 0.8
  Grade 3 redness at injection site | 0 | 0
  Any swelling/induration at injection site | 9.2 | 8.3
  Grade 3 swelling/induration at injection site | 0 | 0
  Any tenderness at injection site | 30.8 | 42.5
  Grade 3 tenderness at injection site | 0 | 0
  Any bruising at injection site | 5.0 | 4.2
  Grade 3 bruising at injection site | 0 | 0

18. Secondary Outcome: Duration of Solicited Local AEs After the First Vaccination
Description: Solicited AEs included AEs that were specifically sought for.
Time Frame: From Day 0 to Day 6 after the first vaccination and up to Day 20 after the first vaccination if AE is ongoing at Day 7
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 120
days
  Pain at injection site | 1.96 (2.423) | 1.67 (1.240)
  Redness at injection site | 1.00 (NA) — Only one participant experienced redness at the injection site so the standard deviation cannot be derived | 1.00 (NA) — Only one participant experienced redness at the injection site so the standard deviation cannot be derived
  Swelling/induration at injection site | 1.64 (0.809) | 2.70 (2.263)
  Tenderness at injection site | 2.24 (1.862) | 1.88 (1.078)
  Bruising at injection site | 5.83 (6.113) | 4.40 (7.057)

19. Secondary Outcome: Frequency and Intensity of Solicited Local AEs After the Second Vaccination
Description: as for outcome 17
Time Frame: From Day 0 to Day 6 after the second vaccination
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 119 | 119
percentage of participants
  Any local solicited AE | 28.6 | 42.9
  Any pain at injection site | 11.8 | 16.8
  Grade 3 pain at injection site | 0 | 0
  Any redness at injection site | 1.7 | 2.5
  Grade 3 redness at injection site | 0 | 0
  Any swelling/induration at injection site | 3.4 | 5.9
  Grade 3 swelling/induration at injection site | 0 | 0
  Any tenderness at injection site | 21.8 | 39.5
  Grade 3 tenderness at injection site | 0 | 0
  Any bruising at injection site | 2.5 | 3.4
  Grade 3 bruising at injection site | 0 | 0

20. Secondary Outcome: Duration of Solicited Local AEs After the Second Vaccination
Description: Solicited AEs included AEs that were specifically sought for.
Time Frame: From Day 0 to Day 6 after the second vaccination and up to Day 20 after the second vaccination if AE is ongoing at Day 7
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 119 | 119
days
  Pain at injection site | 1.50 (0.519) | 2.40 (4.430)
  Redness at injection site | 6.00 (5.657) | 1.67 (1.155)
  Swelling/induration at injection site | 1.75 (0.500) | 1.43 (0.787)
  Tenderness at injection site | 1.62 (0.852) | 2.11 (1.521)
  Bruising at injection site | 8.00 (5.196) | 2.00 (0.707)

21. Secondary Outcome: Frequency and Intensity of Solicited Systemic AEs After the First Vaccination
Description: Solicited AEs included AEs that were specifically sought for. Grade 3 solicited AE definitions: Prevented normal daily activities; Temperature 102.2°F (39.0°C) or more for fevers.
Time Frame: From Day 0 to Day 6 after the first vaccination
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 120
percentage of participants
  Any solicited AE | 37.5 | 53.3
  Any headache | 26.7 | 37.5
  Grade 3 headache | 0 | 0
  Any malaise/feeling generally unwell | 11.7 | 22.5
  Grade 3 Malaise/feeling generally unwell | 0.8 | 0
  Any muscle ache (myalgia) | 15.8 | 19.2
  Grade 3 muscle ache (myalgia) | 0.8 | 0
  Any nausea | 5.8 | 8.3
  Grade 3 nausea | 0.8 | 0.8
  Any chills | 0.8 | 12.5
  Grade 3 chills | 0 | 0
  Any vomiting | 0 | 1.7
  Grade 3 vomiting | 0 | 0
  Any fever | 5.0 | 3.3
  Grade 3 fever | 0 | 0

22. Secondary Outcome: Duration of Solicited Systemic AEs After the First Vaccination
Description: Solicited AEs included AEs that were specifically sought for.
Time Frame: From Day 0 to Day 6 after the first vaccination and up to Day 20 after the first vaccination if AE is ongoing at Day 7
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 120
days
  Headache | 1.15 (0.432) | 1.64 (1.419)
  Malaise/feeling generally unwell | 2.00 (1.328) | 1.47 (1.134)
  Muscle ache (myalgia) | 2.24 (1.729) | 1.67 (1.240)
  Nausea | 1.25 (0.707) | 1.64 (1.286)
  Chills | 3.00 (NA) — Only 1 participant experienced chills so the standard deviation cannot be derived. | 1.38 (0.885)
  Vomiting | NA (NA) — No participants in the CSL425 (15 mcg) group experienced vomiting after the first vaccination. | 2.00 (1.414)
  Fever | 1.14 (0.378) | 1.00 (0.000)

23. Secondary Outcome: Frequency and Intensity of Solicited Systemic AEs After the Second Vaccination
Description: as for outcome 21
Time Frame: From Day 0 to Day 6 after the second vaccination
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 119 | 119
percentage of participants
  Any solicited AE | 19.3 | 32.8
  Any headache | 12.6 | 21.8
  Grade 3 headache | 0 | 0
  Any malaise/feeling generally unwell | 9.2 | 15.1
  Grade 3 Malaise/feeling generally unwell | 0.8 | 0
  Any muscle ache (myalgia) | 9.2 | 11.8
  Grade 3 muscle ache (myalgia) | 0 | 0.8
  Any nausea | 1.7 | 4.2
  Grade 3 nausea | 0 | 0
  Any chills | 0.8 | 1.7
  Grade 3 chills | 0 | 0
  Any vomiting | 0 | 0
  Grade 3 vomiting | 0 | 0
  Any fever | 0 | 2.5
  Grade 3 fever | 0 | 0

24. Secondary Outcome: Duration of Solicited Systemic AEs After the Second Vaccination
Description: Solicited AEs included AEs that were specifically sought for.
Time Frame: as for outcome 20
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 119 | 119
days
  Headache | 1.19 (0.403) | 1.58 (1.173)
  Malaise/feeling generally unwell | 1.64 (0.929) | 2.10 (1.841)
  Muscle ache (myalgia) | 2.08 (2.275) | 2.06 (1.611)
  Nausea | 2.00 (1.414) | 1.29 (0.488)
  Chills | 2.00 (NA) — Only 1 participant experienced chills so the standard deviation cannot be derived. | 1.25 (0.500)
  Vomiting | NA (NA) — No participants in the CSL425 (15 mcg) group experienced vomiting after the second vaccination. | NA (NA) — No participants in the CSL425 (30 mcg) group experienced vomiting after the second vaccination.
  Fever | NA (NA) — No participants in the CSL425 (15 mcg) group experienced fever after the second vaccination. | 1.33 (0.577)

25. Secondary Outcome: Incidence of Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), and New Onset of Chronic Illnesses (NOCIs)
Description: An AESI was defined as an AE for which the association with seasonal influenza vaccine was unclear. A NOCI was defined as the diagnosis of a new medical condition that was chronic in nature, including those potentially controllable by medication (eg, diabetes, asthma).
Time Frame: Up to 180 days after the last vaccination
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 120
percentage of participants
  At least one SAE | 0.8 | 0
  Related SAE | 0 | 0
  At least one AESI | 0 | 0
  Related AESI | 0 | 0
  At least one NOCI | 2.5 | 2.5
  Related NOCI | 0.8 | 1.7

26. Secondary Outcome: Frequency and Intensity of Unsolicited AEs
Description: Unsolicited AEs included AEs other than those specifically sought for.
  The grading definitions were:
  Mild (Grade 1): Symptoms were easily tolerated and did not interfere with daily activities.
  Moderate (Grade 2): Enough discomfort to cause some interference with daily activities.
  Severe (Grade 3): Incapacitating, with inability to work or do usual activities.
Time Frame: From Day 0 to Day 20 after vaccination; up to 180 days after the last vaccination for SAEs, AESIs, and NOCIs
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Number analyzed (Participants) | 120 | 120
percentage of participants
  All unsolicited AEs after the first dose | 40.0 | 35.0
  Grade 1 unsolicited AEs after the first dose | 24.2 | 15.8
  Grade 2 unsolicited AEs after the first dose | 15.0 | 15.0
  Grade 3 unsolicited AEs after the first dose | 0.8 | 4.2
  All unsolicited AEs after the second dose (n=119) | 25.2 | 28.6
  Total unsolicited AEs after doses 1 & 2 | 44.2 | 45.8
  Total grade 1 unsolicited AEs after doses 1 & 2 | 25.0 | 20.8
  Total grade 2 unsolicited AEs after doses 1 & 2 | 17.5 | 20.0
  Total grade 3 unsolicited AEs after doses 1 & 2 | 1.7 | 5.0

ADVERSE EVENTS:
Time Frame: For SAEs: up to 180 days after the last vaccination. For Other AEs: solicited AEs: from Day 0 to Day 6 after each vaccination; unsolicited AEs: from Day 0 to Day 20 after each vaccination; up to 180 days after the last vaccination for AESIs and NOCIs.
Description: Unsolicited AEs presented in the organ system "General disorders" with a footnote of "MedDRA 12.1", were collected under the MedDRA System Organ Class (SOC) 'General disorders and administration site conditions'. Solicited AEs are presented in the organ system "General disorders" and were not collected under the MedDRA SOC.
Arm/Group | CSL425 (15 mcg) | CSL425 (30 mcg)
Serious Adverse Events (participants affected / at risk) | 1/120 | 0/120
Other Adverse Events (participants affected / at risk) | 97/120 | 99/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL425 (15 mcg) (N=120) | CSL425 (30 mcg) (N=120)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSL425 (15 mcg) (N=120) | CSL425 (30 mcg) (N=120)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 4 (8) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 20 (35) | 25 (44)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 9 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (7)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 2 (3)
Toothache (Gastrointestinal disorders) | 3 (5) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 7 (9)
Fatigue (General disorders) | 2 (2) | 3 (3)
Pyrexia (General disorders) | 4 (5) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Pain at injection site (General disorders) | 31 (39) | 36 (47)
Redness at injection site (General disorders) | 3 (3) | 4 (4)
Swelling/Induration at injection site (General disorders) | 13 (15) | 15 (17)
Tenderness at injection site (General disorders) | 47 (63) | 66 (99)
Bruising at injection site (General disorders) | 8 (9) | 9 (10)
Headache (General disorders) | 42 (55) | 52 (87)
Malaise/feeling generally unwell (General disorders) | 22 (32) | 37 (55)
Muscle ache (myalgia) (General disorders) | 26 (33) | 29 (43)
Nausea (General disorders) | 9 (10) | 12 (18)
Chills (General disorders) | 2 (2) | 16 (20)
Vomiting (General disorders) | 0 (0) | 2 (2)
Fever (General disorders) | 6 (7) | 6 (7)
Tooth infection (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
CSL agreements and restrictions on publishing may vary with individual investigators; however, CSL will not prohibit any investigator from publishing. CSL supports the publication of results from all centers of a multi-center trial and generally requires that reports based on single-site data not precede the primary publication of the entire clinical trial.